CLINICAL TRIAL: NCT01687959
Title: Prospective Randomized Clinical Study for Timing of Laparoscopic Cholecystectomy After Endoscopic Retrograde Cholangiography for Acute Biliary Pancreatitis
Brief Title: Timing of Laparoscopic Cholecystectomy After Endoscopic Retrograde Cholangiography for Acute Biliary Pancreatitis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Mustafa Hasbahceci, MD, general surgeon, Bezmialem Vakif University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: BEZM-LC-postERCP
Record Dates: First submitted 2012-09-14; First posted 2012-09-19 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Cholelithiasis Associated With Common Bile Duct Stones
Keywords: cholelithiasis; laparoscopic cholecystectomy; endoscopic sphincterotomy; choledocholithiasis
MeSH Terms: conditions — Cholelithiasis; Choledocholithiasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- activity of peritoneal fibrinolysis (Active Comparator): measurements of peritoneal fibrinolysis using tissue-type plasminogen activator and its specific activity, urokinase-type plasminogen activator, and plasminogen activator inhibitor type 1
  Interventions: Other: tissue sampling from peritoneum of the gallbladder
- surgical outcomes (Active Comparator): surgical outcomes of laparoscopic cholecystectomy
  Interventions: Other: tissue sampling from peritoneum of the gallbladder

INTERVENTIONS:
Other: tissue sampling from peritoneum of the gallbladder — tissue sampling from peritoneum of the gallbladder during laparoscopic cholecystectomy after an acute attack of acute biliary pancreatitis

SUMMARY:
Timing of laparoscopic cholecystectomy following after endoscopic retrograde cholangiography for acute biliary pancreatitis is a controversial issue. There are still many confounding findings offering either early laparoscopic cholecystectomy within 72 hours following endoscopic sphincterotomy or delayed surgery after 6 weeks. Peritoneal plasmin system is known to be an important factor in peritoneal healing and adhesion formation. Measurement of tissue concentrations of tissue-type plasminogen activator and its specific activity, urokinase-type plasminogen activator, and plasminogen activator inhibitor type 1 are thought to be helpful to show peritoneal adhesions after endoscopic sphincterotomy.

DETAILED DESCRIPTION:
Peritoneal fibrinolysis is crucial in peritoneal healing processes and subsequent adhesion formation. It is expected that endoscopic retrograde cholangiography is a trauma causing adhesions around the hepatobiliary area. Such adhesions may cause some difficulty for consequent gallbladder surgery. For that reason, tissue measurements of factors indicating degree of peritoneal healing and adhesion is helpful for timing of such surgical interventions.

Patients are going to be randomized to early and delayed surgery groups. Sampling of peritoneum around the gallbladder during laparoscopic cholecystectomy in patients after endoscopic retrograde cholangiography is performed. Tissue concentrations of tissue-type plasminogen activator and its specific activity, urokinase-type plasminogen activator, and plasminogen activator inhibitor type 1 are going to be studied by using commercial assays.

Peritoneal fibrinolytic activity and surgical outcomes are going to be compared.

ELIGIBILITY:
Inclusion Criteria:

* cholelithiasis following endoscopic retrograde cholangiography for acute biliary pancreatitis

Exclusion Criteria:

* contraindication to laparoscopy
* unsuccessful endoscopic retrograde cholangiography
* complicated acute biliary pancreatitis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-09; Primary Completion 2015-06 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
measurement of peritoneal fibrinolytic response following endoscopic retrograde cholangiography | six months
  measurement of tissue concentrations of tissue-type plasminogen activator and its specific activity, urokinase-type plasminogen activator , and plasminogen activator inhibitor type 1

SECONDARY OUTCOMES:
surgical outcomes of laparoscopic cholecystectomy following endoscopic retrograde cholangiography | six months
  evaluation of surgical outcomes including operating time, morbidity and mortality of laparoscopic cholecystectomy

CONTACTS AND LOCATIONS:
Locations (1):
- department of general surgery; Bezmialem vakif university, Istanbul, Turkey (Türkiye)